CLINICAL TRIAL: NCT02651714
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Tradipitant in Treatment-resistant Pruritus Associated With Atopic Dermatitis
Brief Title: Tradipitant in Treatment-resistant Pruritus Associated With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-2102; NCT02672410 (obsolete NCT alias)
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis
Keywords: eczema; chronic pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental): Oral
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant
  Arms: Tradipitant
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to be conducted in the United States in subjects with treatment-resistant pruritus diagnosed with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female subjects aged 18 - 65 years (inclusive)
* Diagnosed with atopic dermatitis
* Suffering from chronic pruritus with pruritus being actively present

Exclusion Criteria:

* Chronic pruritus due to condition other than atopic dermatitis (AD)
* Participation in a previous tradipitant (LY686017 or VLY-686) trial
* Anyone affiliated with the site or sponsor and/or anyone who may consent under duress
* Any other sound medical reason as determined by the Investigator including any condition which may lead to an unfavorable risk-benefit of study participation, may interfere with study compliance or may confound study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Vanda Investigational Site, Encinitas, California
  - Vanda Investigational Site, Encino, California
  - Vanda Investigational Site, Lomita, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Ormond Beach, Florida
  - Vanda Investigational Site, Columbus, Georgia
  - Vanda Investigational Site, Plainfield, Indiana
  - Vanda Investigational Site, Crowley, Louisiana
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, High Point, North Carolina
  - Vanda Investigational Site, Wilmington, North Carolina
  - Vanda Investigational Site, Winston-Salem, North Carolina
  - Vanda Investigational Site, Portland, Oregon
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Johnston, Rhode Island
  - Vanda Investigational Site, Charleston, South Carolina
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Pflugerville, Texas
  - Vanda Investigational Site, San Antonio, Texas
  - Vanda Investigational Site, West Jordan, Utah
  - Vanda Investigational Site, Seattle, Washington
  - Vanda Investigational Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Tradipitant: Oral
  Tradipitant
- Placebo: Oral
  Placebo
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 84 | 84
Completed | 59 | 56
Not Completed | 25 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.05 (13.139) | 39.13 (13.568) | 40.09 (13.350)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 105
  Male | 32 | 31 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 44
  Not Hispanic or Latino | 61 | 63 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 57 | 106
  Black or African American | 24 | 18 | 42
  Asian | 6 | 5 | 11
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84 | 84 | 168
Average Pruritus VAS at Baseline [Mean (Standard Deviation); unit: mm] — Responses were measured on a 100-mm Visual Analogue Scale (VAS), where the left endpoint was marked "no itch" (0 mm) and in the right endpoint was marked "worst imaginable itch" (100 mm).
  mm | 81.3 (10.78) | 80.3 (8.68) | 80.8 (9.77)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Pruritus Symptoms, as Measured by the 24-hour Average Pruritus Visual Analogue Scale (VAS) Score
Description: Responses were measured on a 100-mm Visual Analogue Scale (VAS), where the left endpoint was marked "no itch" (0 mm) and in the right endpoint was marked "worst imaginable itch" (100 mm).
Time Frame: 56 days
Population: All participants randomized (1:1) to placebo or tradipitant.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 59 | 55
score on a scale | -41.5 (3.89) | -35.8 (4.03)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent through study completion (approximately 100 days) regardless of seriousness or relationship to investigational product.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/82
Other Adverse Events (participants affected / at risk) | 4/83 | 9/82
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tradipitant (N=83) | Placebo (N=82)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT02651714/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT02651714/SAP_001.pdf